CLINICAL TRIAL: NCT04647227
Title: Safety of SEVENFACT® for the Treatment of Bleeding Events in Patients With Hemophilia A or B With Inhibitors
Brief Title: SEVENFACT® for Bleeding Events in Hemophilia With Inhibitors
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: American Thrombosis and Hemostasis Network (Network)
Collaborators: LFB USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATHN 16
Record Dates: First submitted 2020-11-23; First posted 2020-11-30 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hemophilia A With Inhibitor; Hemophilia B With Inhibitor
Keywords: Hemophilia A; Hemophilia B; bleeding event; prophylactic treatment
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — Factor VIIa

STUDY DESIGN:
Intervention Model Description: ATHN 16 is a phase IV multi-center, US-centric, open-label, safety study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Hemophilia A and B Cases (Other): SEVENFACT® has been approved for the treatment of bleeding events in individuals with hemophilia A or B with inhibitors. This study is intended to further investigate the safety and tolerability of SEVENFACT in participants with hemophilia A or B with inhibitors in the presence or absence of prophylactic therapies. Dosing will be at the discretion of the attending physician, and each participant will be supplied with the equivalent of nine 75 µg/kg doses, which aligns with the recommended dosing schedule as provided in SEVENFACT's United States Prescribing Information (USPI). In the event of a bleeding episode (BE), the participant will either self-administer the correct dose under the guidance of the treating investigator or the dose will be administered at a treatment facility.
  Interventions: Drug: coagulation factor VIIa [recombinant]-jncw

INTERVENTIONS:
Drug: coagulation factor VIIa [recombinant]-jncw — a transgenically produced, activated, recombinant, human factor VII (rhFVIIa) protein with the brand name of SEVENFACT®. This protein is a clotting factor in the coagulation cascade that is produced in and purified from the milk of transgenic rabbits. SEVENFACT is approved for the treatment and control of bleeding episodes occurring in adults and adolescents (12 years of age and older) with hemophilia A or B with inhibitors.
  Other Names: SEVENFACT

SUMMARY:
Phase IV multi-center, US-centric, open-label, safety study enrolling participants with Hemophilia A or B with inhibitors, 12 years of age and older, who are either on long term prophylactic treatment (e.g., emicizumab) at risk of experiencing a breakthrough bleeding event (BE), or who are not on prophylactic treatment who may need to control a BE.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the safety of SEVENFACT® when used to treat bleeding episodes in participants with Hemophilia A or B with inhibitors either with or without prophylactic treatment

Study Design:

Phase IV multi-center, US-centric, open-label, safety study enrolling participants with Hemophilia A and B with inhibitors12 years of age and older, who are either on long term prophylactic treatment (e.g., emicizumab) at risk of experiencing a breakthrough bleeding event (BE), or who are not on prophylactic treatment who may need to control a BE.

Study Duration:

Participants will be followed longitudinally from the time of enrollment to the end of their participation in the study. The maximal study duration for any participant in the study will be approximately 4 years from the time of enrollment.

Target Accrual:

This is a multi-site study in which it is anticipated approximately 28 to 55 participants will be enrolled. The study will target enrollment of participants with Hemophilia A and B with inhibitors on prophylaxis with FDA-approved therapies. Enrollment will continue until September 30, 2026, or until the time that the 28th participant is enrolled, whichever comes first.

Data Analysis:

Sample Size Determination:

Results from the study (March 19, 2024, data transfer) with 19 participants enrolled and 3 participant discontinuations were used to calculate the annual bleeding rate for participants receiving prophylactic treatment. Adjusted annualized bleeding rate was calculated at 0.58.

Based on these data, up to 28 participants with hemophilia A and B with inhibitors on FDA-approved prophylaxis treatments will be attempted to enroll.

Analysis Populations:

The Safety Analysis Set is defined as all participants who received at least a single dose of SEVENFACT®. All analyses of safety will be performed based on the safety population, and participants will be analyzed according to the dose of SEVENFACT® that they actually received.

Baseline Characteristics:

Baseline characteristics will be summarized using descriptive statistics for continuous variables, and frequencies and percentages for categorical variables.

Safety Evaluations:

All Adverse Events (AEs) will be graded for severity utilizing Common Terminology Criteria for Adverse Events (CTCAE) v5.0 and coded using Medical Dictionary of Regulatory Activities (MedDRA) version 23.x. The number and percentage of participants with treatment-emergent AEs (TEAEs), serious AEs (SAEs), serious TEAEs and treatment related TEAEs (i.e., adverse drug reactions [ADRs]) will be presented for all participants.

The number of TEAEs, as well as the number and percentage of participants with TEAEs, serious TEAEs, and treatment-related TEAEs will be presented by MedDRA System Organ Class (SOC) and preferred term for all participants.

The number and percentage of participants with treatment-emergent adverse event and/or allergic and anaphylactic reactions will be presented for all participants.

Efficacy Evaluations:

There are no pre-specified efficacy endpoints.

Interim Analysis:

An interim analysis will be conducted after 20 participants have been enrolled into the study. The analysis will seek to characterize baseline, disease, dosing and safety outcome profiles of participants treated with SEVENFACT.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of hemophilia A or B with inhibitors.
2. Be 12 years of age and older
3. Be capable of understanding and willing to comply with the conditions of the protocol or have a legal guardian who is capable of understanding and complying with the conditions of the protocol
4. Have read, understood, and documented written informed consent/assent
5. Be able to provide medical evidence through prior medical history of previous inhibitor levels
6. Be willing and able to use the ATHN mobile application or a paper diary to document BEs and medication usage

Exclusion Criteria:

1. Have a disorder of hemostasis in addition to Hemophilia A or B
2. Have a known or suspected intolerance or hypersensitivity to SEVENFACT® or its ingredients
3. Have a known allergy or hypersensitivity to rabbits or rabbit proteins
4. Are receiving prophylactic treatment for bleeding with a drug or biologic that is not approved for this use by the FDA
5. Have had implantation of an investigational medical device within the prior 6 months
6. Have received an investigational drug within 30 days of the baseline visit
7. Have an elective surgical procedure planned during the duration of their participation in the study*
8. Have any life-threatening disease, or other disease or condition which, in the investigator's judgment, could pose a potential hazard to the patient or interfere with study participation or study outcome (e.g., a history of non responsiveness to bypassing products or thromboembolic disease)

   * Should a participant require an unplanned surgery, the participant will not be withdrawn from the study unless the investigator deems it necessary. Instead, the participant will receive standard of care treatment as determined by the attending physician. If the participant is not withdrawn from the study, the participant's participation in the study will be paused until the investigator feels it is safe for them to continue.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants and percentage of Safety Events (AEs) | From time of consent through BE onset until 3 days after last dose of SEVENFACT®.
  Adverse Events and SAEs defined by the European Haemophilia Safety Surveillance System 2018 (EUHASS) and Serious Adverse Events (SAEs) as defined by the US Food and Drug Association.

CONTACTS AND LOCATIONS:
Overall Officials: Tammuella Chrisentery-Singleton, MD, Principal Investigator — American Thrombosis and Hemostasis Network; Mark Reding, MD, Principal Investigator — University of Minnesota
Locations (21):
- United States (21):
  - Arizona Hemophilia and Thrombosis Center at Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Center for Bleeding Disorders, Little Rock, Arkansas
  - Orthopaedic Institute for Children, Los Angeles, California
  - University of California at Davis UC Davis Hemostasis and Thrombosis Center, Sacramento, California
  - Children's National Hemophilia Center, Washington D.C., District of Columbia
  - Arnold Palmer Hospital for Children - The Haley Center for Children's Cancer and Blood Disorders, Orlando, Florida
  - Hemophilia of Georgia Center for Bleeding and Clotting Disorders of Emory, Adult Division, Atlanta, Georgia
  - Willett Children's Hospital at Memorial University Medical Center, Savannah, Georgia
  - Massachusetts General Hospital Comprehensive Hemophilia and Thrombosis Treatment Center, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - MSU Center for Bleeding and Clotting Disorders, Lansing, Michigan
  - Center for Bleeding and Clotting Disorders, University of Minnesota, Minneapolis, Minnesota
  - Mayo Comprehensive Hemophilia Center, Rochester, Minnesota
  - Kansas City Regional Hemophilia Center, Kansas City, Missouri
  - Northwell Health, Long Island Jewish, New Hyde Park, New York
  - Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - University Hospitals Health System Cleveland, Cleveland, Ohio
  - Oklahoma Center for Bleeding and Clotting Disorders, Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Gulf States Hemophilia and Thrombophilia Center-University of Texas Health Science Center @Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No